CLINICAL TRIAL: NCT03468452
Title: Early Versus Late Extubation After Thymectomy in Patients With Myasthenia Gravis: A Retrospective Analysis
Brief Title: Early Versus Late Extubation in Myasthenia Gravis Patients
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, GengLong Liu, Principal Investigator, First Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: Timing of Extubation
Record Dates: First submitted 2018-03-09; First posted 2018-03-16 (Actual); Last update posted 2018-03-16 (Actual); Status verified 2018-03

CONDITIONS: Myasthenia Gravis Associated With Thymoma
MeSH Terms: interventions — Airway Extubation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Early extubation: The endotracheal tube is removed in the operation room, and no suction support is required after surgery.
  Interventions: Other: extubation
- late extubation: Take the tracheal tube back to the ward for respiratory support or removal of air.
  The catheter is inserted again within 48h.
  Interventions: Other: extubation

INTERVENTIONS:
Other: extubation — Time of extubation

SUMMARY:
MYASTHENIA GRAVIS (MG) is an autoimmune disease characterized by varying degrees of muscle weakness and fatigability worsened with exertion and relieved with rest。Thymectomy plays an important role in the management of these patients because a consistent association between myasthenic and thymic pathology has been recognized.The need for prolonged mechanical ventilation in these patients after thymectomy is determined by their preoperative condition and various perioperative risk factors. Leventhal et al proposed a preoperative scoring system to predict the need for postoperative mechanical ventilation in myasthenic patients undergoing thymectomy based on the following 4 criteria: duration of MG, chronic respiratory disease, dose of pyridostigmine, and vital capacity. However, some investigators discovered that the Leventhal criteria may not be the sole benchmark and that other criteria such as severity of myasthenia,history of myasthenic crisis, and presence of thymoma may be more important in predicting the necessity for prolonged mechanical ventilation after thymectomy. Naguib et al described multivariate determinants of the need for postoperative ventilation after thymectomy in MG patients predominantly on the basis of pulmonary function tests. In addition, the prevalence and presentation of MG may be variable among different ethnic groups. However, there are very few large studies investigating the determinants of prolonged mechanical ventilation after thymectomy. The authors describe the parameters associated with prolonged mechanical ventilation after trans-sternal thymectomy at their institution.

DETAILED DESCRIPTION:
Perioperative variables collected from the patient records were demographic data, duration of the disease,severity of the disease based on Osserman's classification, antiacetylcholine receptor (AChR) antibody positivity, preoperative drug therapy, history of preoperative myasthenic crisis, technique of anesthesia, drugs used for anesthesia, perioperative complications, and duration of postoperative mechanical ventilation. Even though the MG classification by the Myasthenia Gravis Foundation of America is widely accepted,disease severity was graded according to the Osserman and Genkins classification preoperatively as per the authors' institutional protocol.

ELIGIBILITY:
Inclusion Criteria:

* myasthenia gravis patients after thymectomy

Exclusion Criteria:

* not extubation

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: after thymectomy in patients with myasthenia gravis
Sampling Method: Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-11-21 (Actual); Study Completion 2017-12-11 (Actual)

PRIMARY OUTCOMES:
Length of ICU stay | through study completion, an average of 1 year
  Record the time spent in hospital for each patient

CONTACTS AND LOCATIONS:
Overall Officials: Zhenguang Chen, Study Chair — First Affiliated Hospital, Sun Yat-Sen University

IPD SHARING:
Plan to Share IPD: No